CLINICAL TRIAL: NCT06213168
Title: Impact on Mortality of a Strategy Including Continuous Positive Airway Pressure Plus High Flow Nasal Cannula Oxygen Therapy Versus High Flow Nasal Cannula Oxygen Therapy Alone in Patients With de Novo Acute Hypoxemic Respiratory Failure: a Prospective, Randomized Controlled Trial
Acronym: HighCPAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP220813
Record Dates: First submitted 2023-12-18; First posted 2024-01-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-01

CONDITIONS: De Novo Hypoxemic Acute Respiratory Failure (hARF)
Keywords: Continuous positive airway pressure; High flow nasal cannula oxygen therapy; De novo hypoxemic acute respiratory failure; Intensive care unit; Mortality; Mechanical ventilation; Non-invasive ventilation
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: This is a prospective multicentre open-label randomized controlled superiority trial with two parallel arms comparing two oxygenation strategies, HFNC plus CPAP versus HFNC alone, in patients admitted in ICU for de novo hARF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Experimental): Patients assigned to the control group will be continuously treated by HFNC. HFNC will be initiated within one hour following randomization.
  Interventions: Other: HFNC
- HFNC with CPAP (Experimental): Patients assigned to the intervention group will receive high flow nasal oxygen plus CPAP sessions
  Interventions: Other: HFNC; Other: CPAP and HFNC

INTERVENTIONS:
Other: HFNC — Patients assigned to the control group will be continuously treated by HFNC. HFNC will be initiated within one hour following randomization
  Other Names: High flow nasal cannula oxygen therapy
Other: CPAP and HFNC — Patients assigned to the intervention group will receive high flow nasal oxygen plus CPAP sessions
  Other Names: Continuous positive airway pressure and High flow nasal canulae
  Arms: HFNC with CPAP

SUMMARY:
De novo hypoxemic acute respiratory failure (hARF) is one of the main causes of intensive care unit (ICU) admission. In de novo hARF, intubation is associated with a dramatic increase in mortality rate. Compared to standard oxygen, the use of high-flow oxygen nasal cannula (HFNC) might be beneficial to prevent intubation and mortality, although the results of trials and meta-analyses are conflicting. Even with HFNC, the intubation rate remains high. This is the reason why adjunctive therapies, administered in addition to HFNC are needed.

Continuous positive airway pressure (CPAP) is one of these adjunctive therapies. CPAP provides high level of positive end-expiratory pressure that ensures lung recruitment, but without adding inspiratory pressure support, which prevents ventilator induced lung injury. In addition, as opposed to pressure support, CPAP is well tolerated during long periods of time. Therefore, applying CPAP in addition to HFNC may reduce intubation rate and in turn mortality rate.

The present trial will evaluate the impact on mortality of a strategy including continuous positive airway pressure plus high flow nasal cannula oxygen therapy versus high flow nasal cannula oxygen therapy alone in patients with de novo acute hypoxemic respiratory failure: a Prospective, Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years old)
2. Admitted in the ICU for ≤ 24 hours
3. De novo hARF defined by the three following criteria:

   1. Respiratory rate > 25 breaths/min or signs of respiratory distress such as labored breathing or paradoxical inspiration
   2. PaO2/FiO2 ≤ 200 mmHg under HFNC with flow ≥ 45 L/min, actual FiO2 being considered.
   3. Uni or bilateral pulmonary infiltrate on chest X-ray or CT scan
4. Informed consent from the patient or her/his next of kin or another substitute decision maker, or inclusion procedure in emergency if the patient is unable to consent

Exclusion Criteria:

1. Refusal of study participation by the patient or the proxy
2. Anatomical factors precluding the use of a nasal cannula or CPAP
3. Long term oxygen
4. Home CPAP or NIV
5. Hypercapnia indicating NIV (PaCO2 > 45 mmHg)
6. Isolated cardiogenic pulmonary oedema indicating NIV
7. Known pregnancy or breastfeeding
8. Absence of coverage by the French statutory health care insurance system
9. Surgery within the last 6 days
10. Use of vasopressors (norepinephrine>0.3 mcg/kg/min)
11. Glasgow coma scale < 13
12. Urgent need for endotracheal intubation
13. Patients at an end-of-life stage receiving compational oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  Time to death within the 90 days after randomization

SECONDARY OUTCOMES:
Time from randomization to intubation. | 28 days
Intensity of dyspnea until intubation as assessed by a visual analogic scale from zero (no dyspnea) to 100 (maximum possible dyspnea). | 2, 6, 12 and 24 hours
Respiratory rate | 6, 12 and 24 hours
ROX index | 6, 12 and 24 hours
Evaluation of intolerance to oxygenation technique until intubation | 12 and 24 hours
  evaluation based on the following physical criteria: eyes dryness, nose dryness and/or feeling of gastric distention
Discomfort associated with the interface as assessed by a visual analogic scale from zero (no discomfort) to 100 (maximum possible discomfort). | 12 and 24 hours
Level of oxygenation assessed by blood gas that will be sampled on the request of the physician in charge (clinical purpose only). | First 24 hours or until intubation
Use of NIV for one of the following predefined indication criteria. | through study completion
  1. the constitution of a clear indication such as acute-on-chronic respiratory failure with respiratory acidosis (pH < 7.35) or acute cardiogenic pulmonary edema,
  2. pre oxygenation before intubation,
  3. fiberoptic bronchoscopy.
Death within the ICU | through patient participation period,180 days maximum
Time to death | through patient participation period, an average of 180 days maximum
Death within the hospital and time to death. | through patient participation period,180 days maximum
Number of invasive ventilation-free days at 28 days defined as days alive and without intubation. | Between day 1 and day 28
  One point will be given for each day during the measurement period, i.e. from the first day of randomization to day 28 that patients will be both alive and free of invasive mechanical ventilation. Zero value will be given for patients who die before day 28.
Number of HFNC-free days at 28 days defined as days non-intubated, alive and without HFNC. | Between day 1 and day 28.
  One point will be given for each day during the measurement period, i.e. from the first day of randomization to day 28 that patients will be both alive and free of HFNO and invasive mechanical ventilation. Zero value will be given for patients who die or are intubated before day 28.
ICU length of stay. | through patient participation period,180 days maximum
Hospital length of stay. | through patient participation period,180 days maximum
Occurrence of any adverse event during the ICU stay, with a particular focus on hospital or ventilator associated pneumonia, non-respiratory infections, cardiac arrhythmia, and cardiac arrest. | through patient participation period,180 days maximum

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.